CLINICAL TRIAL: NCT05949788
Title: Analyses of Anemia Risk Factors and Prognosis in VLBW Infants.
Brief Title: Analyses of Anemia in Very Low Birth Weight (VLBW) Infants.
Status: Completed | Type: Observational
Sponsor: Shenzhen Bao'an Maternal and Child Health Hospital (Other)
Collaborators: Longhua Hospital Of Baoan District, Shenzhen (Other)
Responsible Party: Principal Investigator, Jun Luo, Principal Investigator, Shenzhen Bao'an Maternal and Child Health Hospital
Other Study IDs: ShenzhenBMCHH
Record Dates: First submitted 2023-07-03; First posted 2023-07-18 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Very Preterm Maturity of Infant; The Risk Factors for Improving the Prognosis of VLBW Infants
Keywords: VLBW; anemia; risk factors; prognosis
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anemia group: The very low birth weight (VLBW) infants meet the diagnostic criteria of neonatal anemia during hospitalization between January 2020 and January 2023.
  Interventions: Other: No intervention
- Control group: The very low birth weight (VLBW) infants are included without anemia during hospitalization between January 2020 and January 2023.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospect study, no direct intervention

SUMMARY:
To study and analyze the association of the severity of anemia with neonatal morbidity and the risk factors of anemia in ealry life (less than 3 days of life) among the very low birth weight (VLBW) infants.

DETAILED DESCRIPTION:
The rescue treatment of very low birth weight (VLBW) infants is the main task of our neonatal intensive care unit (NICU) is this era. Anemia of prematurity (AOP) is one of the most common complication of these infants, which can affect their growth, intelligence, behavior, immunity and hemodynamics, and even endanger their lives in severe situation. It is of great significance to investigate the association of the severity of anemia with neonatal morbidity and the risk factors of anemia in ealry life for improving the prognosis of these infants.

Patient Registry procedures: First, the list of VLBW infants was obtained through medical record search, and sent to the principal investigator (PI) at each center when an infant was eligible for enrollment. Second, patients are included in this study according to the exclusion criteria by PI. Finally, the PI at each center will be responsible for the accuracy,completeness or representativeness of medical records, registry forms,data collection.

Statistical analysis:The two groups were compared by a Χ2-test for categorical variables, Mann-Whitney U Test were used when reporting medians.A P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 32 weeks of gestational age and birth weight below 1500 g and who survive to NICU are eligible for the trial.
* Anemia was defined as a central venous hemoglobin harvested in the first 3 days of life less than two standard deviations below the mean for postnatal age.

Exclusion Criteria:

* Asphyxia (arterial pH <7.0, fifth minute Apgar score <3),
* Twin-to twin-transfusion syndrome,
* Discordant twins (difference in birth weight >20%),
* Major congenital anomalies or chromosomal anomalies,
* Disagree of parents.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All the preterm infants less than 32 weeks of gestational age and birth weight below 1500 g and who survive to neonatal intensive care unit (NICU) are eligible for the trial between January 2020 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Luo, M.D., Study Director — Shenzhen Bao'an Maternal and Child Health Hospital
Locations (1):
- Shenzhen Bao'an Maternal and Child Health Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The outcomes of this study, including the risk factors of anemia in different periods of hospitalization and the influence of anemia in different degrees on prognosis among the very low birth weight (VLBW) infants.

REFERENCES:
- [Background] Everhart KC, Donevant SB, Iskersky VN, Wirth MD, Dail RB. Case Comparison of Preterm Infant Stability During Packed Red Blood Cell Transfusions. Nurs Res. 2023 Jul-Aug 01;72(4):301-309. doi: 10.1097/NNR.0000000000000658. PMID 37350698
- [Background] Patel RM, Knezevic A, Shenvi N, Hinkes M, Keene S, Roback JD, Easley KA, Josephson CD. Association of Red Blood Cell Transfusion, Anemia, and Necrotizing Enterocolitis in Very Low-Birth-Weight Infants. JAMA. 2016 Mar 1;315(9):889-97. doi: 10.1001/jama.2016.1204. PMID 26934258
- [Background] Bellach L, Eigenschink M, Hassanein A, Savran D, Salzer U, Mullner EW, Repa A, Klebermass-Schrehof K, Wisgrill L, Giordano V, Berger A. Packed red blood cell transfusion in preterm infants. Lancet Haematol. 2022 Aug;9(8):e615-e626. doi: 10.1016/S2352-3026(22)00207-1. PMID 35901846
- [Background] Nesterenko TH, Baliga N, Swaintek S, Abdelatif D, Aly H, Mohamed MA. The impact of a multifaceted quality improvement program on the incidence of necrotizing enterocolitis in very low birth weight infants. Pediatr Neonatol. 2022 Mar;63(2):181-187. doi: 10.1016/j.pedneo.2021.10.002. Epub 2021 Dec 5. PMID 34933821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective study on the maternal and infant clinical and electronic records.146 extremely preterm infants with a gestational age of less than 28 weeks were admitted to Bao'an Women's and Children's Hospital affiliated with Jinan University and Longhua District Women's and Children's Hospital from January 1, 2020 to December 31, 2022.
Pre-assignment Details: 45 extremely preterm infants were excluded due to severe birth deformity, twin-twin transfusion syndrome, neonatal hemolytic disease, death within 14 days after birth or transfer to another hospital.
Period: Overall Study
Arm/Group | Anemia Group | Control Group
Started | 36 (March 1, 2023) | 110 (March 1, 2023)
Completed | 25 (March 13, 2024) | 76 (March 13, 2024)
Not Completed | 11 | 34
Not completed — severe birth deformity | 2 | 7
Not completed — twin-twin transfusion syndrome | 2 | 7
Not completed — neonatal hemolytic disease | 3 | 8
Not completed — death within 14 days after birth | 2 | 6
Not completed — transfer to another hospital | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anemia Group | Control Group | Total
Number analyzed (Participants) | 25 | 76 | 101
Age, Continuous [Median (Inter-Quartile Range); unit: weeks (gestational age)] — the median gestational age in anemia group
  weeks (gestational age)
    Gestational age | 26 [24.86 to 26.86] | 26.79 [26 to 27.57] | 26.43 [25.86 to 27.43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 28 | 39
  Male | 14 | 48 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 25 | 76 | 101

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Early Onset Sepsis in VLBW Infants With AOP.
Description: The incidence of early onset sepsis in very low birth weigh (VLBW) infants with anemia of prematurity (AOP)
Time Frame: through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anemia Group | Control Group
Number analyzed (Participants) | 25 | 76
Participants
  Early onset sepsis | 18 | 34
  Non-early onset sepsis | 7 | 42

2. Secondary Outcome: The Maternal Hb Levels Before Birth Among VLBW Infants With AOP.
Description: The maternal hemoglobin (Hb) levels in very low birth weight (VLBW) infants with anemia of prematurity (AOP)
Time Frame: Through study completion, an average of 6 months
Measure: Median (Inter-Quartile Range); unit: g/L
Groups:
- The Anemia Group: The VLBW infants with anemia
- The Non-anemia Group: The VLBW infants without anemia
Arm/Group | The Anemia Group | The Non-anemia Group
Number analyzed (Participants) | 25 | 76
g/L | 111 [94.5 to 120.5] | 107 [97.5 to 119.5]

3. Secondary Outcome: Mortality and Morbidity Among Extremely Preterm Infants With Anemia of Prematurity (AOP)
Description: The incidence of death and morbidity among extremely preterm infants with AOP and without.
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anemia Group | Control Group
Number analyzed (Participants) | 25 | 76
Participants
  moderate or severe BPD | 7 | 20
  ROP (greater than II) | 12 | 39
  NEC | 3 | 6
  neonatal sepsis | 17 | 39
  IVH | 7 | 16
  EUGR | 3 | 14
  Death | 3 | 4

ADVERSE EVENTS:
Time Frame: "through study completion, an average of 6 months"
Description: Two in anemia group and six in non-anemia group were excluded due to death within 14 days after birth.
  Three of 25 patients in anemia group were died, and four of 76 patients in non-anemia group were died.
  In anemia group: Two died from late onset sepsis, another died from necrotizing enterocolitis.
  In non-anemia group: Four died from late onset sepsis.
Arm/Group | Anemia Group | Control Group
All-Cause Mortality (participants affected / at risk) | 5/36 | 10/110
Serious Adverse Events (participants affected / at risk) | 5/36 | 10/110
Other Adverse Events (participants affected / at risk) | 20/36 | 45/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anemia Group (N=36) | Control Group (N=110)
Death (Infections and infestations) | 2 (2) | 6 (6) — In anemia group: Two died from late onset sepsis. In non-anemia group: Six died from late onset sepsis.
Death (Reproductive system and breast disorders) | 2 (2) | 4 (4) — One in anemia group and two in non-anemia group were died from respiratory failure within 14 days after birth.One in anemia group and two in non-anemia group were died from pneumothorax within 14 days after birth.
Death (Gastrointestinal disorders) | 1 (1) | 0 (0) — One in anemia group died from necrotizing enterocolitis.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anemia Group (N=36) | Control Group (N=110)
Neonatal sepsis (Infections and infestations) | 17 (17) | 39 (39) — Neonatal sepsis diagnosis required positive culture along with clinical signs (fever; hypothermia; lethargy; tachypnea; apnea/bradycardia; cyanosis; and hypoglycemia not explained by other diagnoses) or laboratory signs of infection.
NEC (Gastrointestinal disorders) | 3 (3) | 6 (6) — NEC was defined as stage 2 or higher based on Bell's criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05949788/Prot_SAP_002.pdf